CLINICAL TRIAL: NCT05366153
Title: Risk-guided Disease managEment Plan to prevEnt CAD in Patients Treated With Previous Cancer (REDEEM-CAD)
Brief Title: Risk-guided Disease managEment Plan to prevEnt CAD in Patients Treated With Previous Cancer
Acronym: REDEEM-CAD
Status: Recruiting | Type: Observational
Sponsor: Baker Heart and Diabetes Institute (Other)
Collaborators: Western Health, Australia (Other Government); Northern Hospital, Australia (Other); Menzies Institute for Medical Research (Other); Peter MacCallum Cancer Centre, Australia (Other); The Alfred (Other)
Responsible Party: Sponsor
Other Study IDs: 134-22
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Coronary CT scans
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivor Screening/Management Plan: In cancer survivors;
  1. A novel clinical and CT imaging-based screening algorithm to select those most likely to develop coronary artery disease,
  2. A clinical review to ensure optimal risk factor control and cardiac protection.
  Interventions: Diagnostic Test: Coronary CT
- Non-cancer Screening/Management Plan: In matched non-cancer patients (from EDCAD trial);
  1. A novel clinical and CT imaging-based screening algorithm to select those most likely to develop coronary artery disease,
  2. A clinical review to ensure optimal risk factor control and cardiac protection.
  Interventions: Diagnostic Test: Coronary CT

INTERVENTIONS:
Diagnostic Test: Coronary CT — Screening/Management Plan

SUMMARY:
REDEEM-CAD is a prospective multi-centre study of CAD risk evaluation and management in cancer survivors 40-70 years with chemotherapy or radiotherapy >5 years ago.

DETAILED DESCRIPTION:
REDEEM-CAD is a prospective multi-centre study in which a process of evaluating the risk of coronary artery disease is studied in cancer survivors 40-70 years with chemotherapy or radiotherapy >5 years ago. The efficacy of this CAD risk evaluation will be compared with the broad community in two existing studies - CAUGHT-CAD and EDCAD. This unique Screening/Management Plan (SMP) has 2 components; 1) A novel clinical and imaging-based screening algorithm to select those most likely to develop coronary artery disease, 2) A clinical review to ensure optimal risk factor control and cardio protection.

Follow-up of treated patients will continue for an average of 36 months, with clinic reviews at 12, 24 and 36 months. The results will define the prevalence of subclinical coronary artery disease, and the feasibility and the efficacy of the SMP.

ELIGIBILITY:
Inclusion Criteria:

A history of cancer >5 y ago associated with potential cardiotoxicity from chemotherapy and/or radiotherapy (chiefly survivors of breast cancer, Hodgkin's lymphoma and prostate cancer).

Exclusion Criteria:

* Unable to provide written informed consent to participate in this study
* Known coronary artery disease at recruitment
* History of previous coronary artery disease
* Inability to acquire interpretable CT images
* Contraindications/Intolerance to or already taking statin therapy
* Oncologic (or other) life expectancy <12 months or any other medical condition (including pregnancy) that results in the belief (deemed by the Chief Investigators) that it is not appropriate for the patient to participate in this trial

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer survivors 40-70 years with chemotherapy or radiotherapy >5 years ago
Sampling Method: Non-Probability Sample
Enrollment: 748 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of evaluated patients who should undergo CAD prevention | 3 years
  High clinical risk, or intermediate risk with CAC score >0

SECONDARY OUTCOMES:
Proportion with critical CAD | 3 years
  Coronary stenosis >70% by CT coronary angiogram
Proportion at intermediate clinical risk | 3 years
  Intermediate clinical risk (0.8-2.0% annualized risk by Pooled Cohort Equation)
Statin responsiveness | 3 year follow-up
  Change in plaque volume

CONTACTS AND LOCATIONS:
Overall Officials: Tom Marwick, MBBS,PhD,MPH, Principal Investigator — Baker Heart and Diabetes Institute
Locations (2):
- Australia (2):
  - Tom Marwick, Hobart, Tasmania
  - Baker Heart and Diabetes Institute, Melbourne, Victoria

REFERENCES:
- [Derived] Soh CH, Smith J, Shrestha S, Nolan M, Wong J, Nerlekar N, Marwick TH. Screening for coronary artery disease among cancer survivors: rationale and design of the REDEEM-CAD study. Cardiooncology. 2025 Feb 4;11(1):10. doi: 10.1186/s40959-025-00308-7. PMID 39905553